CLINICAL TRIAL: NCT05380336
Title: Medico-economic Evaluation Comparing the Impact of the New Fixed-dose Nivolumab Regimen With the Old mg/kg Regimen in the Management of Patients With Metastatic Cancer
Acronym: IMEPOCA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0371
Record Dates: First submitted 2022-05-05; First posted 2022-05-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Cancer
Keywords: nivolumab; lung; kidney cancer; melanoma; cost-effectiveness
MeSH Terms: conditions — Neoplasm Metastasis; Kidney Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with the Nivolumab weight-dependent dosage: Patients treated for their metastatic cancer with Nivolumab, with a dosage calculated upon their weight (3mg/kg every two weeks).
- Patients with the Nivolumab fixed dosage: Patients treated for their metastatic cancer with Nivolumab, with a fixed-dose regimen of 240 mg every 2 weeks or 480 mg every 4 weeks

SUMMARY:
Nivolumab is a selective monoclonal antibody that binds to the Programmed cell Death 1 (PD-1) receptor and causes reduced tumor growth. It is currently approved in France in many indications. The firsts therapeutics indications validated by the French health authorities from 2015 - metastatic melanoma2, squamous and non-squamous NSCLC, Kidney cells carcinoma - were based on clinical trials demonstrating a clinical advantage over standard nivolumab treatment at a dose of 3mg/kg every two weeks.

By comparing the results predicted by simulation based on a pharmacokinetic model with those obtained in clinical trials, the manufacturer of nivolumab concluded that a fixed dose of 240 mg was equivalent to that calculated based on the weight of the patients, and the European and then French health authorities have validated this change in clinical practice The objective of the IMEPOCA study is to assess in real life the economic and clinical impact of the dose modification of nivolumab that occurred in December 2018 in France.

In order to assess the economic efficiency of the change in dose strategy at the national level, 2 cohorts of patients from the National Health Data System (SNDS), treated for metastatic cancer and followed up over 1 year will be compared: one having benefited from the weight-dependent dosage and the other having benefited from the fixed dosage

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic melanoma, non-small cell lung cancer (NSCLC) and renal cell carcinoma treated with nivolumab monotherapy
* Patients whose nivolumab treatment was initiated between 2015 and 2020
* Patients with health insurance

Exclusion Criteria:

* Patients whose nivolumab treatment initiated in 2017 in mg/kg has progressed to a fixed dose in the 1st year of treatment
* Patients treated with nivolumab in the adjuvant setting for melanoma with lymph node involvement or metastatic disease and who have undergone complete resection (Approval in 2018 for this indication)
* Patients whose nivolumab treatment has been initiated in 2018

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients with metastatic cancers treated with nivolumab: lung cancer, melanoma and kidney cancer.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness analysis of the new nivolumab fixed-dose regimen of 240 mg every 2 weeks or 480 mg every 4 weeks compared to the old regimen of 3 mg/kg every 2 weeks in the management of patients with metastatic cancers. | 1 year
  Incremental cost effectiveness ratio (in cost per year of life alive) according to a collective perspective and a time horizon of one year, according to the type of cancer

SECONDARY OUTCOMES:
Comparison of the patients characteristics between the 2015-2017 "de novo" cohort in mg/kg dosage and the 2019-2020 de novo cohort in fixed dosage by type of cancer | baseline
  Initial characteristics of patients treated with nivolumab (age, sex, average weight, medical history, previous treatments)
Comparison of nivolumab length of treatment between the 2015-2017 "de novo" cohort in mg/kg dosage and the 2019-2020 de novo cohort in fixed dosage by type of cancer | 1 year
  treatment time frame, including interruption or suspension periods
Comparison of nivolumab treatment dosage between the 2015-2017 "de novo" cohort in mg/kg dosage and the 2019-2020 de novo cohort in fixed dosage by type of cancer | 1 year
  Average dosage of nivolumab per patient hospitalisation
Comparison of number of hospitalisations for nivolumab treatment between the 2015-2017 "de novo" cohort in mg/kg dosage and the 2019-2020 de novo cohort in fixed dosage by type of cancer | 1 year
  Average number of hospitalisations for nivolumab treatment, per patient
Comparison of complications related to nivolumab between the 2015-2017 "de novo" cohort in mg/kg dosage and the 2019-2020 de novo cohort in fixed dosage by type of cancer | 1 year
  number of complications related to nivolumab, identified through the health care consumptions
Patient survival analysis | 6 years
  patients date of death, by cancer type
Duration of treatment response | 6 years
  Duration of treatment
Budget impact analysis of the nivolumab fixed-dose regimen of 240 mg every 2 weeks or 480 mg every 4 weeks compared to the old regimen of 3 mg/kg every 2 weeks | 7 years (2015-2022)
  Comparison of the costs of nivolumab fixed-dose regimen of 240 mg every 2 weeks or 480 mg every 4 weeks compared to the old regimen of 3 mg/kg every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CORMIER, MD, Principal Investigator — Nantes University Hospital